CLINICAL TRIAL: NCT06545526
Title: The Chemopreventive Effect of Celecoxib Monotherapy Versus Combination of Celecoxib and Metformin in Patients With Familial Adenomatous Polyposis: a Pilot Randomized, Open-label, Comparative Study
Brief Title: Chemopreventive Effect of Combination of Celecoxib and Metformin in Patients With Familial Adenomatous Polyposis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2024-0371
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- celecoxib monotherapy (Active Comparator): celecoxib [400mg, twice a day] for 6 months
  Interventions: Drug: celecoxib monotherapy
- celecoxib and metformin combination (Experimental): celecoxib [400mg, twice a day] and metformin [1g, twice a day] for 6 months
  Interventions: Drug: celecoxib and metformin combination

INTERVENTIONS:
Drug: celecoxib monotherapy — Patients will be randomly assigned in a 1:1 ratio to receive celecoxib monotherapy or combination of celecoxib and metformin orally for 6 months: celecoxib [400mg, twice a day] in arm 1, celecoxib [400mg, twice a day] and metformin [1g, twice a day] in arm 2.
  Arms: celecoxib monotherapy
Drug: celecoxib and metformin combination — Patients will be randomly assigned in a 1:1 ratio to receive celecoxib monotherapy or combination of celecoxib and metformin orally for 6 months: celecoxib [400mg, twice a day] in arm 1, celecoxib [400mg, twice a day] and metformin [1g, twice a day] in arm 2.
  Arms: celecoxib and metformin combination

SUMMARY:
Familial adenomatous polyposis (FAP) leads to adenomas and eventual adenocarcinomas in colon and less frequently, duodenum. Chemopreventive strategies have been studied in FAP patients to delay the development of adenomas and cancers. The non-steroidal anti-inflammatory drugs (NSAIDs) and selective cyclooxygenase-2 inhibitor have shown the regression of colorectal and duodenal adenomas in FAP patients. However, these drugs showed gastrointestinal damage and cardiovascular risks, and new preventive strategies are needed. Metformin, an anti-diabetic drug, has recently been suggested to have a suppressive effect on tumorigenesis via inhibition of mTOR pathway, and have an inhibitory effect on polyp recurrence after removal of sporadic colorectal polyps. In addition, metformin has a number of potential mechnisms of carciovascular bebefit. We devised a randomized, open-label, comparative study to evaluate the effect of combination of celecoxib and metformin on polyps of colorectum and duodenum in FAP patients.

DETAILED DESCRIPTION:
This clinical trial is a randomized, open-label, comparative study to evaluate the effect of combination of celecoxib and metformin on polyps of colorectum and duodenum in FAP patients. FAP patients, satisfied an enrollment criteria, will be randomly assigned in a 1:1 ratio to receive celecoxib monotherapy or combination of celecoxib and metformin orally for 6 months. The base-line and six-month endoscopic examination (colonoscopy/sigmoidoscopy and upper gastrointestinal endoscopy) will be recorded, and photographs will be taken at the tattoo-marked area. The number and size of polyps, and a qualitative assessment of the total extent of polyposis will be measured.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with familial adenomatous polyposis(FAP) who are 20 to 55 years of age.

2. FAP patients who have colonic or duodenal polyp. 3. FAP patients who have five or more polyps 2mm or more in diameter in endoscopic examination.

Exclusion Criteria:

* 1. FAP patients who had a history of colectomy within the previous 12 months or need to undergo colectomy within 8 months after randomization.

  2. FAP patients with malignant disease, including colorectal cancer. 3. FAP patients who used NSAIDs (non-steroidal anti-inflammatory drugs) or aspirin three or more times a week within 3 months of randomization.

  4. Pregnant or breast-feeding patients. 5. Patients with cardiovascular diseases, peptic ulcer diseases and diabetes. 6. Patients with abnormal results of serum laboratory tests (renal function and liver function test).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change of the number and size of polyps in colon and/or duodenum. | After six-month administration of celecoxib monotherapy or combination of celecoxib and metformin
  At the base-line endoscopy (colonoscopy and upper gastrointestinal endoscopy), india-ink tattoo will be placed in the ascending colon, sigmoid colon/rectum, and duodenum. In case of patient with retained rectum after colectomy and ileorectal anastomosis, sigmoidoscopy will be peformed. The base-line and six-month endoscopic examination will be recorded, and photographs will be taken at the tattoo-marked area and used for measurements of the number and size of polyps. The diameter of a polyp will be measured with the aid of biopsy forceps included in the photographic field, and only distinct polyps at least 2 mm in diameter will be counted.

SECONDARY OUTCOMES:
A qualitative assessment of the total extent of colorectal and duodenal polyposis | After six-month administration of celecoxib monotherapy or combination of celecoxib and metformin
  A qualitative assessment of the total extent of colorectal polyposis will be conducted via video review(at base line and month 6) by two endoscopists experienced in the management of FAP, and scored as the same as, better than, or worse than base-line endoscopic findings, without the endoscopists' being aware of treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea